CLINICAL TRIAL: NCT06440889
Title: Prospective, Open-Label, Control-group, Proof-Of-Science, Real-life Setting, Clinical Safety and Efficacy Study of a Bio-Ray Knee Guard in Panelists with Varicose Vein and Self-Declared Knee Pain.
Brief Title: A Clinical Study to Determine the Safety and Efficacy of Bio-Ray Knee Guard in Panelists with Varicose Vein and Knee Pain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NovoBliss Research Pvt Ltd (Other)
Collaborators: Winnox Cosmeceutics Sdn. Bhd (Industry)
Responsible Party: Principal Investigator, Dr Nayan Patel, Sub-Investigator, NovoBliss Research Pvt Ltd
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NB240023-WU
Record Dates: First submitted 2024-05-27; First posted 2024-06-04 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Varicose Veins with Self-declared Knee Pain

STUDY DESIGN:
Intervention Model Description: Prospective, Open-Label, Control-group, Proof-Of-Science, Real-life Setting, Clinical Safety and Efficacy Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Varicose Vein Group (Experimental): Ebene Bio-Ray Knee Guard Wear the test product in the daytime for about 1-2 hours. Then, proceed to gradually lengthen the duration of wear to 4-6 and 6-8 hours.
  Interventions: Device: Bio-Ray Knee Guard
- Healthy Group (Other): Ebene Bio-Ray Knee Guard Wear the test product in the daytime for about 1-2 hours. Then, proceed to gradually lengthen the duration of wear to 4-6 and 6-8 hours.
  Interventions: Device: Bio-Ray Knee Guard

INTERVENTIONS:
Device: Bio-Ray Knee Guard — Wear the metal guard (test product) for 1-2 hours during the first week, and then for 6-8 hours thereafter. (minimum for 4 hours)

SUMMARY:
Prospective, Open-Label, Control-group, Proof-Of-Science, Real-life Setting Clinical Safety and Efficacy Study of a Bio-Ray Knee Guard in Panelists with varicose vein and Self-Declared Knee Pain.

Sample size for this proof-of-science study is kept 32 panelists aged 35 to 70 years with self-declared knee pain and varicose veins will be enrolled and 32 healthy panelists will be enrolled.

DETAILED DESCRIPTION:
Potential panelists will undergo screening based on predefined inclusion and exclusion criteria only after obtaining written informed consent.

Panelists shall be instructed to visit the facility for the following scheduled visits:

Visit 01 (Day 01): Screening, enrolment, evaluations at baseline, test product and *subject diary distribution, followed by evaluations after 1 hour (+10 minutes).

Visit 02 (Day 03 +1 day): Evaluations at Day 03 (+1 day).

Visit 03 (07 ±2 days): 1-week evaluations at Day 07 (±2 days).

Visit 04 (28±2 days): Subject diary review, followed by end of study evaluations.

ELIGIBILITY:
Inclusion Criteria:

1. Panelists of either gender, aged from 35 to 70 years (both inclusive) at the time of informed consent.
2. Non-pregnant and non-lactating adult females having a self-reported negative urine pregnancy test.
3. Panelist of childbearing potential, is practicing and agrees to maintain an established method of birth control (IUD, hormonal implant device/injection, regular use of birth control pills or patch, diaphragm, condoms with spermicide or sponge with spermicidal jelly, cream or foam, vasectomy or abstinence).
4. 32 panelists with clinical diagnosis of varicose veins in any of the leg with C2 class as per CEAP classification (Appendix II), with self-declared knee pain.
5. 32 healthy panelists will be enrolled.
6. Documented written informed consent from the panelists.
7. Panelists having willingness and ability to adhere to study directions, and agreeing not to use any other or wear any other similar product at the same designated site for this study and returning for all specified visits for follow-up.
8. Panelists are currently not enrolled in an active investigational study or have participated in similar investigational study within 30 days prior to enrolment.

Exclusion Criteria:

1. Any significant or serious cardiovascular, pulmonary, hepatic, renal, gastrointestinal, haematological, endocrinological, metabolic, neurological or psychiatric disease which, in the opinion of the PI, renders the panelists unfit to take part in the study.
2. Any recent surgery which may hinder in the study specific assessments and overall outcome.
3. Panelists with class C3 to C6 of CEAP classification.
4. Panelists who are currently on medication therapy for varicose veins, deep vein thrombosis or chronic venous insufficiency.
5. Panelists taking or have taken medication(s) which, in the Investigator's judgment, make them ineligible or places them at undue risk.
6. Panelists are currently enrolled in an active investigational study or have participated in an investigational study within 30 days prior to enrolment.
7. Females who are pregnant or breastfeeding or planning to become pregnant during the study period.
8. Panelists who are not willing to adhere to the study protocol.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2024-05-31 (Actual); Primary Completion 2024-10-04 (Actual); Study Completion 2024-10-04 (Actual)

PRIMARY OUTCOMES:
Change in Blood Parameters (D-dimer) | On Day 01 (Baseline) before usage and at Day 28 (±2 days) of test product usage, within group and between group.
  To assess the effectiveness of the test product in terms of determining the biomarker D-dimer.
Change in Blood Parameters (C-reactive protein) | On Day 01 (Baseline) before usage and at Day 28 (±2 days) of test product usage, within group and between group.
  To assess the effectiveness of the test product in terms of determining the biomarker C-reactive protein.
Change in Blood Parameters (Rheumatoid factor) | On Day 01 (Baseline) before usage and at Day 28 (±2 days) of test product usage, within group and between group.
  To assess the effectiveness of the test product in terms of determining the biomarker rheumatoid factor.
Change in Blood Parameters (anti-CCP antibodies) | On Day 01 (Baseline) before usage and at Day 28 (±2 days) of test product usage, within group and between group.
  To assess the effectiveness of the test product in terms of determining the biomarker anti-CCP antibodies.
Change in Blood Parameters (MCP-1) | On Day 01 (Baseline) before usage and at Day 28 (±2 days) of test product usage, within group and between group.
  To assess the effectiveness of the test product in terms of determining the biomarker MCP-1.
Change in Blood Parameters (IL-6) | On Day 01 (Baseline) before usage and at Day 28 (±2 days) of test product usage, within group and between group.
  To assess the effectiveness of the test product in terms of determining the biomarker IL-6.
Change in Blood Parameters (TNF-α) | On Day 01 (Baseline) before usage and at Day 28 (±2 days) of test product usage, within group and between group.
  To assess the effectiveness of the test product in terms of determining the biomarker TNF-α.
Change in Blood Circulation (SFJ) | On Day 01 (Baseline) before usage and at Day 28 (±2 days) of test product usage, within group and between group.
  To assess the effectiveness of the test product in terms of change in blood circulation of saphenofemoral junction by duplex ultrasound.
Change in Blood Circulation (GSV) | On Day 01 (Baseline) before usage and at Day 28 (±2 days) of test product usage, within group and between group.
  To assess the effectiveness of the test product in terms of change in blood circulation of great saphenous vein by duplex ultrasound.
Change in Blood Circulation (SSV) | On Day 01 (Baseline) before usage and at Day 28 (±2 days) of test product usage, within group and between group.
  To assess the effectiveness of the test product in terms of change in blood circulation of small saphenous veins by duplex ultrasound.
Change in blood valve function (SFJ) | On Day 01 (Baseline) before usage and at Day 28 (±2 days) of test product usage, within group and between group.
  To assess the effectiveness of the test product in terms of change in blood valve function of saphenofemoral junction by duplex ultrasound.
Change in blood valve function (GSV) | On Day 01 (Baseline) before usage and at Day 28 (±2 days) of test product usage, within group and between group.
  To assess the effectiveness of the test product in terms of change in blood valve function of great saphenous vein by duplex ultrasound.
Change in blood valve function (SSV) | On Day 01 (Baseline) before usage and at Day 28 (±2 days) of test product usage, within group and between group.
  To assess the effectiveness of the test product in terms of change in blood valve function of small saphenous vein by duplex ultrasound.
Change in vessel anatomy (SFJ) | On Day 01 (Baseline) before usage and at Day 28 (±2 days) of test product usage, within group and between group.
  To assess the effectiveness of the test product in terms of change in vessel anatomy of saphenofemoral junction by duplex ultrasound.
Change in vessel anatomy (GSV) | On Day 01 (Baseline) before usage and at Day 28 (±2 days) of test product usage, within group and between group.
  To assess the effectiveness of the test product in terms of change in vessel anatomy of great saphenous vein by duplex ultrasound.
Change in vessel anatomy (SSV) | On Day 01 (Baseline) before usage and at Day 28 (±2 days) of test product usage, within group and between group.
  To assess the effectiveness of the test product in terms of change in vessel anatomy of small saphenous vein by duplex ultrasound.
Change in overall health of knee joint. | On Day 01 (Baseline) before usage, at 1-hour (+10 minutes), Day 03 (+1 days), Day 07 (±2 days) and Day 28 (±2 days) of test product usage.
  To assess the effectiveness of the test product in terms of change in overall health of knee joint based on questionnaire.
Change in VAS pain score (only for vericose vain panelist) | On Day 01 (Baseline) before usage, at 1-hour (+10 minutes), Day 03 (+1 days), Day 07 (±2 days) and Day 28 (±2 days) of test product usage.
  To assess the effectiveness of the test product in terms of change in VAS pain score of Knee. Where 0= No pain 10 = worst pain
Change in CEAP classification (Clinical-Etiology-Anatomy-Pathophysiology) | On Day 01 (Baseline) before usage, at 1-hour (+10 minutes), Day 03 (+1 days), Day 07 (±2 days) and Day 28 (±2 days) of test product usage.
  To assess effectiveness of the test product in terms of change in CEAP classification of the severity of varicose vein. C0 = No visible or palpable signs of venous disease, C1= Telangiectasias or reticular veins C2 = Varicose vein and

SECONDARY OUTCOMES:
Change in blood pressure | On Day 01 (Baseline) before usage, at 1-hour (+10 minutes), Day 03 (+1 days), Day 07 (±2 days) and Day 28 (±2 days) of test product usage, within group and between group.
  To assess the effectiveness of the test product in terms of change in blood pressure of upper leg (standing or sitting).
Change in blood pressure | On Day 01 (Baseline) before usage, at 1-hour (+10 minutes), Day 03 (+1 days), Day 07 (±2 days) and Day 28 (±2 days) of test product usage, within group and between group.
  To assess the effectiveness of the test product in terms of change in blood pressure of lower leg (standing or sitting).
Change in ankle-brachial index | On Day 01 (Baseline) before usage, at 1-hour (+10 minutes), Day 03 (+1 days), Day 07 (±2 days) and Day 28 (±2 days) of test product usage, within group and between group.
  To assess the effectiveness of the test product in terms of change in ankle-brachial index.
Change in body leg temperature | On Day 01 (Baseline) before usage, at 1-hour (+10 minutes), Day 03 (+1 days), Day 07 (±2 days) and Day 28 (±2 days) of test product usage, within group and between group.
  To assess the effectiveness of the test product in terms of change in body leg temperature by Infrared camera (thermal image).
Overall improvement in symptoms and satisfaction with the use of test product | On Day 01 (Baseline) before usage, at 1-hour (+10 minutes), Day 03 (+1 days), Day 07 (±2 days) and Day 28 (±2 days) of test product usage.
  To assess the effectiveness of the test product in terms of overall improvement in symptoms and satisfaction with the use of test product using subjective perception questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Nayan K Patel K Patel, Principal Investigator — NovoBliss Research Pvt Ltd
Locations (1):
- NovoBliss Research Pvt.Ltd, Ahmedabad, Gujarat, India

IPD SHARING:
Plan to Share IPD: No